CLINICAL TRIAL: NCT02265289
Title: Influence of Oral Doses of 75 mg Clopidogrel on the Pharmacodynamics and Safety of Fradafiban After Oral Doses of 30 mg Lefradafiban Tid Over 8 Days in Healthy Male Subjects. An Intra-individual, Open Trial.
Brief Title: Influence of Clopidogrel on the Pharmacodynamics and Safety of Fradafiban in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 509.302
Record Dates: First submitted 2014-10-14; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — lefradafiban; Clopidogrel

ARMS (1):
- Lefradafiban with clopidogrel (Experimental): All patients received the same treatment:
  * Lefradafiban only (day 1-4)
  * Lefradafiban in combination with Clopidogrel (day 5-8)
  * Clopidogrel only (day 9-12)
  Interventions: Drug: Lefradafiban; Drug: Clopidogrel

INTERVENTIONS:
Drug: Lefradafiban
Drug: Clopidogrel

SUMMARY:
To assess the influence of 75 mg Clopidogrel on the pharmacodynamics and safety of 30 mg Lefradafiban tid

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with good clinical practice (GCP) and local legislation
* Healthy male subjects
* Age ≥ 18 and ≤ 45 years
* Broca ≥ - 20 % and ≤ + 20 %

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of

  * Allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
  * Any bleeding disorder including prolonged or habitual bleeding
  * Other hematologic disease
  * Cerebral bleeding (e.g. after a car accident
  * Commotio cerebri
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during the trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* History of any familial bleeding disorder
* Thrombocytes < 150000/µl

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 1999-01; Primary Completion 1999-02 (Actual)

PRIMARY OUTCOMES:
Inhibition of platelet aggregation in platelet rich plasma (PRP) | Up to 383:30 hours after first drug administration
Fibrinogen receptor occupancy levels (FRO) | Up to 383:30 hours after first drug administration
Maximum concentration of the analyte in plasma at steady state (Cmax) | Up to 383:30 hours after first drug administration
Area under the concentration-time curve of the analyte in plasma (AUC) | Up to 383:30 hours after first drug administration
Amount of the analyte excreted unchanged in the urine (Ae) | Up to 176:00 hours after first drug administration

SECONDARY OUTCOMES:
Number of subjects with adverse events | up to 5 days after last drug administration
Changes from baseline in 12-lead ECG | Pre-dose and 384:30 hours after first drug administration
Number of subjects with clinically significant findings in vital signs | up to 5 days after last drug administration
  systolic and diastolic blood pressure, pulse rate
Changes from baseline in bleeding time | Pre-dose and 384:30 hours after first drug administration